CLINICAL TRIAL: NCT00298038
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy, Safety and Tolerability of Rifaximin 550 mg BID For 6 Months In Preventing Hepatic Encephalopathy
Brief Title: A 6-month Efficacy, Safety, and Tolerability Study of Rifaximin In Preventing Hepatic Encephalopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RFHE3001
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rifaximin (Experimental): Participants were administered a single rifaximin 550 milligram (mg) tablet 2 times per day (approximately every 12 hours) for 6 months or until a breakthrough episode of hepatic encephalopathy or another reason for discontinuation.
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Participants were administered a single matching placebo tablet 2 times per day (approximately every 12 hours) for 6 months or until a breakthrough episode of hepatic encephalopathy or another reason for discontinuation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Oral
  Other Names: Xifaxan®
  Arms: Rifaximin
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the study drug is safe and effective in preventing hepatic encephalopathy (HE).

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent Form
* In remission from past HE
* Uses appropriate birth control measures
* More than or equal to 18 years of age
* Must have potential to benefit from treatment
* Recent prior HE episodes
* Capable and willing to comply with all study procedures
* Participant has personal support available
* Has a certain Model End Stage Liver Disease (MELD) score
* Recent transjugular intrahepatic portosystemic shunt (TIPS) placement or revision

Exclusion Criteria:

* Significant medical conditions, medical conditions that may impact study participation, or Investigator decision not to include
* Allergies to the study drug or similar drugs
* Laboratory abnormalities
* Recent participation in another clinical trial
* History of non-compliance
* Pregnant or at risk of pregnancy, or is lactating
* Recent alcohol consumption
* Active bacterial or viral Infections
* Bowel issues
* Active malignancy
* On a prohibited medication
* Liver transplant expected in near term
* Lactulose intolerance
* Participant shows presence of intestinal obstruction or has inflammatory bowel disease
* Ongoing or recent GI bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2005-12-19 (Actual); Primary Completion 2008-08-15 (Actual); Study Completion 2008-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Companies

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Flamm SL, Mullen KD, Heimanson Z, Sanyal AJ. Rifaximin has the potential to prevent complications of cirrhosis. Therap Adv Gastroenterol. 2018 Sep 28;11:1756284818800307. doi: 10.1177/1756284818800307. eCollection 2018. PMID 30283499
- [Derived] Sanyal A, Younossi ZM, Bass NM, Mullen KD, Poordad F, Brown RS, Vemuru RP, Mazen Jamal M, Huang S, Merchant K, Bortey E, Forbes WP. Randomised clinical trial: rifaximin improves health-related quality of life in cirrhotic patients with hepatic encephalopathy - a double-blind placebo-controlled study. Aliment Pharmacol Ther. 2011 Oct;34(8):853-61. doi: 10.1111/j.1365-2036.2011.04808.x. Epub 2011 Aug 17. PMID 21848797
- [Derived] Bass NM, Mullen KD, Sanyal A, Poordad F, Neff G, Leevy CB, Sigal S, Sheikh MY, Beavers K, Frederick T, Teperman L, Hillebrand D, Huang S, Merchant K, Shaw A, Bortey E, Forbes WP. Rifaximin treatment in hepatic encephalopathy. N Engl J Med. 2010 Mar 25;362(12):1071-81. doi: 10.1056/NEJMoa0907893. PMID 20335583

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were to be withdrawn from the study after experiencing a breakthrough overt hepatic encephalopathy (HE) episode.
Groups:
- Rifaximin: Participants were administered a single rifaximin 550 milligrams (mg) tablet 2 times per day (approximately every 12 hours) for 6 months or until a breakthrough episode of hepatic encephalopathy or another reason for discontinuation.
Period: Overall Study
Arm/Group | Rifaximin | Placebo
Started | 140 | 159
Received At Least 1 Dose Of Study Drug | 140 | 159
Completed | 88 | 66
Not Completed | 52 | 93
Not completed — Lost to Follow-up | 0 | 1
Not completed — Liver Transplant | 0 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Death | 6 | 3
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Adverse Event | 8 | 7
Not completed — Breakthrough overt HE episode | 28 | 69
Not completed — Noncompliance | 1 | 0
Not completed — Cocaine Abuse | 1 | 0
Not completed — Severe Gastrointestinal Bleed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug (ITT population).
Groups:
- Rifaximin: Participants were administered a single rifaximin 550 mg tablet 2 times per day (approximately every 12 hours) for 6 months or until a breakthrough episode of hepatic encephalopathy or another reason for discontinuation.
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Placebo | Total
Number analyzed (Participants) | 140 | 159 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.57) | 56.8 (9.18) | 56.2 (56.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 52 | 117
  Male | 75 | 107 | 182

OUTCOME MEASURES:

1. Primary Outcome: Time To The First Breakthrough Overt HE Episode
Description: Time to a breakthrough overt HE episode was the duration (number of days) from time of first dose of study drug to the first breakthrough overt HE episode. A breakthrough overt HE episode was defined as an increase of Conn score from Grade 0 or 1 to ≥2, or an increase in Conn and asterixis score of 1 grade each for those participants who entered the study with a Conn score of 0. Participants who completed the study and did not experience a breakthrough overt HE episode were censored at the time of their 6-month visit. Participants who terminated early for reasons other than a breakthrough overt HE episode were contacted at 6 months from randomization to determine if they had experienced a breakthrough overt HE event or other outcome. Participants without breakthrough overt HE were censored at the time of last contact or death, whichever was earlier. The number of events of a first breakthrough overt HE episode during the treatment interval is presented.
Time Frame: Baseline up to 6 Months (168 days)
Population: Randomized participants who received at least 1 dose of study drug (ITT population). Assuming censored cases were at risk for half of the interval for onset of breakthrough HE episode, the censored cases only counted for half in figuring number at risk. Numbers at risk were rounded up to whole integers.
Measure: Number; unit: events
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 140 | 159
events
  0 to <28 Days: number analyzed (Participants) | 140 | 158
  0 to <28 Days | 13 | 20
  28 to <56 Days: number analyzed (Participants) | 126 | 137
  28 to <56 Days | 4 | 23
  56 to <84 Days: number analyzed (Participants) | 120 | 113
  56 to <84 Days | 6 | 14
  84 to <140 Days: number analyzed (Participants) | 112 | 98
  84 to <140 Days | 7 | 10
  140 to <168 Days: number analyzed (Participants) | 98 | 84
  140 to <168 Days | 1 | 6
  ≥168 Days: number analyzed (Participants) | 46 | 38
  ≥168 Days | 0 | 0
Statistical Analysis 1: Comparison: Rifaximin vs Placebo; Test type: Superiority — Analysis based on the overall comparison of time to the first breakthrough overt HE episode between rifaximin and placebo groups adjusting for analysis region, using the Cox proportional hazards model (Score test, [that is, Log rank test stratified by analysis region]) with a 2-sided test at a significance level of 0.05 under the proportional hazards assumption; p < 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.421, 95% CI 2-sided [0.276 to 0.641]

2. Secondary Outcome: Time To First HE-related Hospitalization
Description: Time to first HE-related hospitalization is defined as the duration (number of days) between the first dose of study drug and the date of first HE-related hospitalization. Participants who discontinued prior to hospitalization due to HE and prior to completion of the 6-month treatment period were censored at the time of discontinuation. The number of participants with their first HE-related hospitalization per interval is presented. The number of events of the first HE-related hospitalization during the treatment interval is presented.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 140 | 159
events
  0 to <28 Days: number analyzed (Participants) | 139 | 155
  0 to <28 Days | 4 | 11
  28 to <56 Days: number analyzed (Participants) | 130 | 132
  28 to <56 Days | 4 | 12
  56 to <84 Days: number analyzed (Participants) | 119 | 108
  56 to <84 Days | 4 | 7
  84 to 140 Days: number analyzed (Participants) | 106 | 88
  84 to 140 Days | 5 | 4
  140 to <168 Days: number analyzed (Participants) | 92 | 72
  140 to <168 Days | 2 | 2
  ≥168 Days: number analyzed (Participants) | 43 | 34
  ≥168 Days | 0 | 0

3. Secondary Outcome: Time To Any Increase From Baseline In Conn Score
Description: Time to any increase in Conn score (mental state grade) was computed as the number of days from the first dose of study drug to the initial occurrence of an increase from baseline in Conn score. Conn score range: Grade 0 (no behavioral abnormality) to Grade 4 (coma; unable to test mental state). Participants who discontinued prior to experiencing an increase in Conn score and prior to completion of the 6-month treatment period were censored at the time of discontinuation. The number of events of the initial occurrence of an increase from baseline in Conn score during the treatment interval is presented.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 140 | 159
events
  0 to <28 Days: number analyzed (Participants) | 139 | 156
  0 to <28 Days | 17 | 26
  28 to <56 Days: number analyzed (Participants) | 119 | 125
  28 to <56 Days | 5 | 21
  56 to <84 Days: number analyzed (Participants) | 109 | 100
  56 to <84 Days | 9 | 15
  84 to <140 Days: number analyzed (Participants) | 94 | 80
  84 to <140 Days | 5 | 10
  140 to <168 Days: number analyzed (Participants) | 79 | 62
  140 to <168 Days | 0 | 5
  ≥168 Days: number analyzed (Participants) | 37 | 27
  ≥168 Days | 1 | 0

4. Secondary Outcome: Time To Any Increase From Baseline In Asterixis Grade
Description: Time to any increase in asterixis grade was computed as the number of days from the first dose of study drug to the initial occurrence of an increase from baseline in asterixis grade. Asterixis (flapping tremor) was determined with the participant holding both arms and forearms extended with wrists dorsiflexed and fingers open for ≥30 seconds per standard practice. Asterixis grade range: Grade 0 (no abnormal movement) to Grade 4 (almost continuous flapping motions). Participants who discontinued prior to experiencing an increase in asterixis grade and prior to completion of the 6-month treatment period were censored at the time of discontinuation. The number of events of the initial occurrence of an increase from baseline in asterixis grade during the treatment interval is presented.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 140 | 159
events
  0 to <28 Days: number analyzed (Participants) | 137 | 154
  0 to <28 Days | 13 | 20
  28 to <56 Days: number analyzed (Participants) | 116 | 120
  28 to <56 Days | 7 | 15
  56 to <84 Days: number analyzed (Participants) | 101 | 91
  56 to <84 Days | 7 | 4
  84 to <140 Days: number analyzed (Participants) | 87 | 76
  84 to <140 Days | 3 | 6
  140 to <168 Days: number analyzed (Participants) | 74 | 61
  140 to <168 Days | 1 | 4
  ≥168 Days: number analyzed (Participants) | 34 | 27
  ≥168 Days | 1 | 1

5. Secondary Outcome: Mean Change From Baseline In Fatigue Domain Score On The CLDQ At End Of Treatment
Description: The 29-item Chronic Liver Disease Questionnaire (CLDQ) questionnaire consists of the following domains: fatigue, activity, emotional function, abdominal symptoms, systemic symptoms, and worry. Participants ranked their level of fatigue by using a 7-point scale from the worst response (1, high degree of fatigue) to the best response (7, minimal fatigue).
Time Frame: Baseline, 6 months (End Of Treatment)
Population: Randomized participants who received at least 1 dose of study drug (ITT population) and able to complete the questionnaire at the applicable time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 140 | 159
score on a scale
  Baseline: number analyzed (Participants) | 99 | 114
  Baseline | 3.28 (1.326) | 3.34 (1.406)
  Change from Baseline: number analyzed (Participants) | 95 | 105
  Change from Baseline | 0.30 (1.262) | 0.11 (1.319)

6. Secondary Outcome: Mean Change From Baseline In Venous Ammonia Concentration At End Of Treatment
Description: Venous blood samples (10 mL) were collected at Baseline/Randomization (Day 0) and Days 28, 84, and 168. Baseline value was the last available value prior to first dose of study drug, and end of treatment value was the last available post-baseline value during the treatment period.
Time Frame: Baseline, Month 6 (End Of Treatment)
Population: Randomized participants who received at least 1 dose of study drug (ITT population) with evaluable venous ammonia data.
Measure: Mean (Standard Deviation); unit: microgram per deciliter (ug/dL)
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 140 | 159
microgram per deciliter (ug/dL)
  Baseline: number analyzed (Participants) | 132 | 149
  Baseline | 87.9 (47.76) | 92.1 (55.24)
  Change from Baseline: number analyzed (Participants) | 125 | 133
  Change from Baseline | -5.7 (46.77) | -1.2 (60.98)

ADVERSE EVENTS:
Time Frame: Baseline up to 6.5 months
Description: Randomized participants who received at least 1 dose of study drug (ITT population).
Arm/Group | Rifaximin | Placebo
Serious Adverse Events (participants affected / at risk) | 51/140 | 63/159
Other Adverse Events (participants affected / at risk) | 91/140 | 101/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin (N=140) | Placebo (N=159)
Ascites (Gastrointestinal disorders) | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Endophthalmitis (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 | 2
Peritonitis (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Generalised oedema (General disorders) | 3 | 2
Multi-organ failure (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 6
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Liver transplant rejection (Immune system disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 2
Clostridium colitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hepatic neoplasm malignant resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 16 | 34
Syncope (Nervous system disorders) | 2 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respite care (Social circumstances) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin (N=140) | Placebo (N=159)
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 19 | 21
Diarrhoea (Gastrointestinal disorders) | 15 | 21
Ascites (Gastrointestinal disorders) | 15 | 13
Abdominal pain (Gastrointestinal disorders) | 11 | 13
Vomiting (Gastrointestinal disorders) | 8 | 14
Abdominal distension (Gastrointestinal disorders) | 10 | 11
Constipation (Gastrointestinal disorders) | 9 | 9
Abdominal pain upper (Gastrointestinal disorders) | 9 | 8
Pyrexia (General disorders) | 8 | 5
Fatigue (General disorders) | 17 | 18
Oedema peripheral (General disorders) | 21 | 13
Asthenia (General disorders) | 4 | 11
Nasopharyngitis (Infections and infestations) | 10 | 10
Urinary tract infection (Infections and infestations) | 6 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4
Headache (Nervous system disorders) | 14 | 17
Dizziness (Nervous system disorders) | 18 | 12
Insomnia (Psychiatric disorders) | 10 | 11
Depression (Psychiatric disorders) | 10 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 10
Rash (Skin and subcutaneous tissue disorders) | 7 | 6
Hepatic encephalopathy (Nervous system disorders) | 8 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.